CLINICAL TRIAL: NCT03585010
Title: Brain Response Associated With Parent-based Treatment for Childhood Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023649; 4R33MH115113-03 (NIH); 1R61MH115113-01A1 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorder of Childhood; Separation Anxiety Disorder of Childhood; Social Anxiety Disorder of Childhood; Generalized Anxiety Disorder
Keywords: anxiety disorders
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessments will conducted by independent evaluators, blind to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Parenting for Anxious Childhood Emotions (Experimental): Parent-based treatment for childhood anxiety disorders
  Interventions: Behavioral: Supportive Parenting for Anxious Childhood Emotions
- Parent Educational Support or CBT (Active Comparator): Parent-based intervention for childhood anxiety disorders (phase 1) or child based treatment for childhood anxiety disorders (phase 2)
  Interventions: Behavioral: Parent Educational Support; Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Supportive Parenting for Anxious Childhood Emotions — 12 sessions with parents
  Arms: Supportive Parenting for Anxious Childhood Emotions
Behavioral: Parent Educational Support — 12 sessions with parents
  Arms: Parent Educational Support or CBT
Behavioral: Cognitive-Behavioral Therapy — 12 sessions with child
  Arms: Parent Educational Support or CBT

SUMMARY:
This study aims to investigate whether a parent-based treatment for childhood anxiety disorders engages child brain circuitry implicated in children's reliance on parents to reduce anxiety (R61), and whether change in child brain circuitry is associated with reduction in child anxiety (R33).

DETAILED DESCRIPTION:
Specific Aims: Anxiety disorders impact up to one-third of children, cause tremendous suffering, increase risk for psychiatric and medical morbidity, impair school and social functioning, and cost billions of dollars each year. Data consistently show that child anxiety is characterized by amygdala hyperactivity and deficits in prefrontal control of the amygdala. Emerging data link these disruptions to anxious children's over-reliance on parents for amygdala-medial prefrontal cortex (mPFC) engagement and anxiety reduction.

In the first phase of this study we aim to demonstrate that an entirely parent-based psychosocial treatment with no child involvement, Supportive Parenting for Anxious Childhood Emotions (SPACE), engages an amygdala-mPFC target in anxious children, lessening child reliance on parents to reduce amygdala reactivity.

Cross-species neurobiological evidence indicates that parental presence reduces amygdala reactivity and activates the mPFC to reduce offspring anxiety. In humans we recently demonstrated parental presence increases functional connectivity between their child's mPFC and amygdala, reducing the child's amygdala reactivity and anxiety. In a healthy sample, parental engagement of child amygdala-mPFC connectivity was linked to the child's reliance on parents for help with anxiety. Data from clinically anxious children likewise show parental presence engages child mPFC, and data we collected since our previous submission demonstrate that parental presence reduces amygdala reactivity in clinically anxious children.

Offspring's natural reliance on parents for anxiety reduction is magnified in clinically anxious children. Parents become deeply enmeshed in their child's symptoms through the process of family accommodation, defined as change in parents' behavior to help the child avoid or alleviate anxiety. In clinically anxious children, 90% report depending on parents to reduce their anxiety, and 97% of parents report accommodating their anxious child's symptoms. These cross-generational patterns of parental entanglement in their child's anxiety symptoms contribute to the immense burden, distress, and costs of pediatric anxiety (e.g., parents missing work to be with their anxious child). Anxious children's reliance on parents for anxiety reduction may disrupt the child's ability to independently reduce amygdala reactivity and anxiety.

We developed SPACE to translate these neurobiological and clinical research findings into a manualized parent-based treatment focused on reducing family accommodation in parents of anxious children. Preliminary data from a randomized clinical trial show that after 12 weeks of parents receiving SPACE (N=29), with no therapist-child contact, family accommodation and child anxiety were significantly reduced. We propose that SPACE engages anxious children's amygdala-mPFC circuitry, lessening their reliance on parents to reduce amygdala reactivity.

The first phase of the study will examine clinically anxious children's (N=90, 7-10 yrs) amygdala-mPFC response to fear faces when (A) the child's parent is beside them holding their hand during the fMRI scan (Parent-Present), and (B) the child is alone during the scan (Parent-Absent) (within-subjects design). Children with primary separation, social, or generalized anxiety disorder diagnoses, the most common childhood anxiety disorders, will serve as participants. Children will complete Parent-Present and Parent-Absent scans PRE- and POST-SPACE, or PRE- and POST-Parent Educational Support (PES), the comparator treatment that controls for treatment duration and therapist-parent contact. We expect SPACE will lessen child reliance on parental presence to engage amygdala-mPFC circuitry and reduce child amygdala reactivity. Aim 1: Demonstrate SPACE lessens children's reliance on parents to reduce amygdala reactivity (target engagement). Hyp 1: Child reliance on parental presence to reduce amygdala reactivity, (i.e., the difference between child amygdala reactivity in the Parent-Present and Parent-Absent scan), will decrease significantly from PRE- to POST-SPACE, as compared with PRE- to POST-PES. If Hyp 1 is confirmed we will proceed to the the second phase of the study.

The second phase of the study will be performed to re-demonstrate target engagement in SPACE, compared to cognitive-behavioral therapy (CBT); demonstrate target engagement is associated with symptom reduction in SPACE; and demonstrate SPACE's acceptability/feasibility. The second phase will enroll 136 clinically anxious children (7-10 yrs), randomly assigned to SPACE or CBT. Aim 1: Re-demonstrate target engagement in SPACE. Hyp 1: Child reliance on parental presence to reduce amygdala reactivity will decrease significantly from PRE- to POST-SPACE, as compared with PRE- to POST-CBT. Aim 2: Demonstrate target engagement is associated with symptom reduction in SPACE. Hyp 2: Reduction in child anxiety from PRE- to POST-SPACE will be significantly associated with reduction in child reliance on parental presence to reduce amygdala reactivity. Aim 3: Establish acceptability and feasibility of SPACE. Hyp 3: SPACE will be acceptable and feasible to administer, and comparable to CBT. The second phase will also provide insight into the relative efficacy of SPACE, to inform future research and development of SPACE.

This study has the potential to provide groundbreaking results, with major public health impact, on how parent-based treatments can target disrupted neurobiological processes in children with psychopathology. These novel data will inform decision-making about a large-scale study (R01) to confirm the efficacy of SPACE and examine personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal
* Clinical diagnosis of primary anxiety disorder
* Must not have another mental illness more impairing than the most impairing anxiety disorder
* IQ of at least 80.

Exclusion Criteria:

* Neurological disorders (including seizures)
* Organic mental disorders, psychotic disorders, or pervasive developmental disorders
* High likelihood of hurting themselves or others
* Current psychosocial or psychopharmacological treatment
* History of neurological illness or head injury with loss of consciousness > 5 minutes
* Vision or physical disability that interferes with seeing stimuli presented briefly on computer screen and/or clicking a mouse button rapidly and repeatedly
* Contraindications for MRI scanning (e.g., metal implants, pacemakers, braces, claustrophobia, pregnancy, weight > 250 pounds).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | 12 weeks
  The PARS is a clinician-administered measure of anxiety severity in children and adolescents.
  Total scores on PARS are used as indicator of anxiety severity. Total scores range from 0-35, with higher scores indicating more severe anxiety.

SECONDARY OUTCOMES:
Multimodal Anxiety Scale for Children (MASC) | 12 weeks
  The MASC is a self-report measure of anxiety severity, completed by children and parents separately.
  MASC generates a total anxiety score and several sub scales:
  Total scores: range from 0-150 Separation/Phobias scores: range from 0-27 Generalized anxiety scores: range from 0-30 Social anxiety scores: range from 0-27 Obsessive-compulsive symptom scores: 0-50 Physical symptoms scores: 0-60 For Total score and all sub-scales, higher scores indicate more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Eli R Lebowitz, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for primary and secondary measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available six months after study completion
Access Criteria: Data access requests will be reviewed by review panel and requestors will sign a Data Access Agreement

DOCUMENTS (1):
  • Informed Consent Form (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT03585010/ICF_000.pdf